CLINICAL TRIAL: NCT01527604
Title: Effects of Avenanthramide-enriched Oats on Inflammation in Obese Adults With Central Adiposity: A Randomized Clinical Trial
Brief Title: Effects of Avenanthramide-enriched Oats on Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB9930
Record Dates: First submitted 2012-01-30; First posted 2012-02-07 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Avenanthramide-enriched oat muffin (Active Comparator)
  Interventions: Other: Avenanthramide-enriched oats
- Refined flour muffin (Placebo Comparator)
  Interventions: Other: Refined flour absent avenanthramides

INTERVENTIONS:
Other: Avenanthramide-enriched oats — avenanthramide-enriched oats, delivered as muffins at a dose of 2 muffins per day for 56 days.
  Arms: Avenanthramide-enriched oat muffin
Other: Refined flour absent avenanthramides — refined flour absent avenanthramides, delivered as muffins at a dose of 2 muffins per day for 56 days.
  Arms: Refined flour muffin

SUMMARY:
The objective of this randomized, double-blinded, placebo-controlled, parallel trial is to determine whether consuming avenanthramide-enriched oats daily for 8 weeks on can improve biomarkers of inflammation in older, obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Men & postmenopausal women, age 50 years and over
* BMI 30-36 kg/m2
* waist:hip ratio > 0.8 for women, > 0.9 for men

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* Individuals taking estrogen
* Use of cholesterol-lowering medications
* Use of blood pressure-lowering medications
* Regular use of any stomach acid-lowering medications, laxatives (including fiber supplements) or anti-diarrheal medications(prescription or over-the-counter [OTC])
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 95 mmHg
* Regular use of oral steroids
* Regular daily intake of ≥ 2 alcoholic drinks
* Strict vegetarians
* No dietary supplements, including those containing any vitamins, minerals, herbs, plant concentrates (including garlic, gingko, St. John's wort) homeopathic remedies, probiotics, or fish oil (including cod liver oil), for one month prior to study admission

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers of inflammation compared with placebo | Baseline and 8 weeks
  Primary outcome measures will include selected biomarkers of inflammation in blood, i.e., pro-inflammatory cytokines, chemokines, as well as other inflammatory markers (i.e., high sensitivity C-reactive protein).

SECONDARY OUTCOMES:
Change in biomarkers of glucoregulation, plasma lipids, and blood pressure compared with placebo | Baseline and 8 weeks
  Secondary outcomes will include plasma markers of glucoregulation (fasting glucose, insulin, HOMA), plasma lipids (total cholesterol, HDL, LDL, triglycerides), and blood pressure (BP).

CONTACTS AND LOCATIONS:
Overall Officials: Diane L. McKay, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States